CLINICAL TRIAL: NCT00853385
Title: Phase 3 Randomized, Double-Blind, Active Comparator, Placebo-Controlled Study Of The Efficacy And Safety Of 2 Doses Of CP 690,550 In Patients With Active Rheumatoid Arthritis On Background Methotrexate
Brief Title: A Phase 3 Study Comparing 2 Doses Of CP-690,550 And The Active Comparator, Humira (Adalimumab) Vs. Placebo For Treatment Of Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921064
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis
Keywords: oral DMARD; JAK inhibitor; clinical trial
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 5mg (Experimental)
  Interventions: Drug: CP 690,550
- 10 mg (Experimental)
  Interventions: Drug: CP-690,550
- Placebo Sequence 1 (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo Sequence 2 (Placebo Comparator)
  Interventions: Other: Placebo
- adalimumab (Active Comparator)
  Interventions: Biological: Biologic TNFi

INTERVENTIONS:
Drug: CP 690,550 — tablets 5 mg BID PO plus q2 week placebo SC injections for 12 months
  Arms: 5mg
Drug: CP-690,550 — tablets 10 mg BID PO plus q2 week placebo SC injections for 12 months
  Arms: 10 mg
Other: Placebo — placebo tablets BID PO advance to 5mg CP 690,550 BID at Month 3 or 6 visit plus q2 week placebo SC injections for 12 months
  Arms: Placebo Sequence 1
Other: Placebo — tablets BID PO advance tablets to10mg CP 690,550 BID at Month 3 or 6 visit plus q2 week placebo SC injections for 12 months
  Arms: Placebo Sequence 2
Biological: Biologic TNFi — placebo tablets BID PO plus adalimumab 40 mg q2 week SC injections for 12 months
  Other Names: Humira (Adalimumab)
  Arms: adalimumab

SUMMARY:
This is a comparative study of CP 690,550, Humira (adalimumab) and placebo on background methotrexate in patients with Rheumatoid Arthritis. The study is intended to provide evidence of the efficacy and safety of CP 690,550 when dosed 5 mg and 10 mg twice a day on background methotrexate in adult patients with moderate to severe Rheumatoid Arthritis. It is intended to confirm the benefits of CP-690,550 in improving signs and symptoms and physical function that were observed in Rheumatoid Arthritis. An active comparator, adalimumab, is also included.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of RA based upon the American College of Rheumatology (ACR) 1987 Revised Criteria.
* The patient must have had an inadequate response to methotrexate and have active disease, as defined by both: ≥6 joints tender or painful on motion; and ≥6 joints swollen; and fulfills 1 of the following 2 criteria at Screening: 1.ESR (Westergren method) >28 mm in the local laboratory. 2. CRP >7 mg/L in the central laboratory.
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis.
* The patient must have been on a stable dose of 7.5 mg to 25 mg weekly of methotrexate and washed out of all other DMARDs.

Exclusion Criteria:

* Blood dyscrasias including confirmed: 1. Hemoglobin <9 g/dL or Hematocrit <30%; 2. White blood cell count <3,000 cu.mm. Absolute neutrophil count <1,200 cu.mm; 4. Platelet count <100,000/L
* History of any other autoimmune rheumatic disease other than Sjogren's syndrome
* No malignancy or history of malignancy.
* History of infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator, within the 6 months prior to the first dose of study drug
* Patients who have failed any TNFi for either lack of efficacy or a TNFi mechanism related adverse event.
* Patients who have previously received adalimumab therapy for any reason.
* Patients who are contraindicated for treatment with adalimumab in accordance with the approved local label.
* Patients meeting the New York Heart Association Class III and Class IV Congestive Heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (113):
- United States (36):
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Paradise Valley, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Fair Oaks, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Largo, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Pinellas Park, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Haverhill, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lubbock, Texas
  - Pfizer Investigational Site, Mesquite, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Clarksburg, West Virginia
- Australia (4):
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Cairns, Queensland
  - Pfizer Investigational Site, Maroochydore, Queensland
  - Pfizer Investigational Site, Malvern East, Victoria
- Pfizer Investigational Site, Sarajevo, Bosnia and Herzegovina
- Bulgaria (4):
  - Pfizer Investigational Site, Pleven
  - Pfizer Investigational Site, Plovdiv
  - Pfizer Investigational Site, Sevlievo
  - Pfizer Investigational Site, Sofia
- Canada (8):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Lunenburg, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Trois-Rivières, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Chile (3):
  - Pfizer Investigational Site, Rancagua, Región del Libertador General Bernardo O’Higgins
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Providencia, Santiago, RM
- Costa Rica (2):
  - Pfizer Investigational Site, Cartago, Cartago Province
  - Pfizer Investigational Site, San José, Provincia de San José
- Croatia (3):
  - Pfizer Investigational Site, Osijek
  - Pfizer Investigational Site, Split
  - Pfizer Investigational Site, Zagreb
- Czechia (7):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Brno-Židenice
  - Pfizer Investigational Site, Hlučín
  - Pfizer Investigational Site, Pardubice
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha 11 - Chodov
  - Pfizer Investigational Site, Zlín
- Denmark (2):
  - Pfizer Investigational Site, Frederiksberg
  - Pfizer Investigational Site, Randers NOE
- Pfizer Investigational Site, Santo Domingo, Santo Domingo Province, Dominican Republic
- Pfizer Investigational Site, Hyvinkää, Finland
- Germany (7):
  - Pfizer Investigational Site, Aachen
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Herne
  - Pfizer Investigational Site, Ratingen
  - Pfizer Investigational Site, Würzburg
- Mexico (4):
  - Pfizer Investigational Site, Guadalajara, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Morelia, Michoacán
  - Pfizer Investigational Site, San Luis Potosí City, San Luis Potosí
- Philippines (3):
  - Pfizer Investigational Site, Lipa City, Batangas
  - Pfizer Investigational Site, Angeles City, Pampanga
  - Pfizer Investigational Site, Cebu City
- Poland (7):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Cieszyn
  - Pfizer Investigational Site, Kościan
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Sopot
  - Pfizer Investigational Site, Torun
  - Pfizer Investigational Site, Warsaw
- Slovakia (6):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Dunajská Streda
  - Pfizer Investigational Site, Košice
  - Pfizer Investigational Site, Nové Zámky
  - Pfizer Investigational Site, Povazska Dystrica
  - Pfizer Investigational Site, Žilina
- South Korea (3):
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Gwangju
  - Pfizer Investigational Site, Seoul
- Spain (6):
  - Pfizer Investigational Site, A Coruña, A Coruña
  - Pfizer Investigational Site, Santiago de Compostela, A Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Vigo, Pontevedra
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
- Thailand (2):
  - Pfizer Investigational Site, Rajathevee, Bangkok
  - Pfizer Investigational Site, Amphoe Muang, Chiang Mai
- United Kingdom (3):
  - Pfizer Investigational Site, Metropolitan Borough of Wirral, Merseyside
  - Pfizer Investigational Site, Cannock, Staffs
  - Pfizer Investigational Site, Dudley, West Midlands

REFERENCES:
- [Derived] Strand V, Schulze-Koops H, Al-Emadi S, Kinch CD, Gruben D, Germino R, Connell CA, Mysler E. Sex differences in the efficacy, safety and persistence of tofacitinib in patients with rheumatoid arthritis: a post hoc analysis of phase III and long-term extension trials. BMJ Open. 2025 Dec 24;15(12):e082366. doi: 10.1136/bmjopen-2023-082366. PMID 41448717
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Citera G, Jain R, Irazoque F, Madariaga H, Gruben D, Wang L, Stockert L, Santana K, Ebrahim A, Ponce de Leon D. Tofacitinib Efficacy in Patients with Rheumatoid Arthritis and Probable Depression/Anxiety: Post Hoc Analysis of Phase 3 and 3b/4 Randomized Controlled Trials. Rheumatol Ther. 2024 Feb;11(1):35-50. doi: 10.1007/s40744-023-00612-7. Epub 2023 Nov 5. PMID 37925660
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Dougados M, Taylor PC, Bingham CO 3rd, Fallon L, Brault Y, Roychoudhury S, Wang L, Kessouri M. The effect of tofacitinib on residual pain in patients with rheumatoid arthritis and psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002478. doi: 10.1136/rmdopen-2022-002478. PMID 36814062
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Dikranian AH, Gonzalez-Gay MA, Wellborne F, Alvaro-Gracia JM, Takiya L, Stockert L, Paulissen J, Shi H, Tatulych S, Curtis JR. Efficacy of tofacitinib in patients with rheumatoid arthritis stratified by baseline body mass index: an analysis of pooled data from phase 3 studies. RMD Open. 2022 May;8(1):e002103. doi: 10.1136/rmdopen-2021-002103. PMID 35577477
- [Derived] Bartlett SJ, Bingham CO, van Vollenhoven R, Murray C, Gruben D, Gold DA, Cella D. The impact of tofacitinib on fatigue, sleep, and health-related quality of life in patients with rheumatoid arthritis: a post hoc analysis of data from Phase 3 trials. Arthritis Res Ther. 2022 Apr 5;24(1):83. doi: 10.1186/s13075-022-02724-x. PMID 35382883
- [Derived] Dikranian A, Gold D, Bessette L, Nash P, Azevedo VF, Wang L, Woolcott J, Shapiro AB, Szumski A, Fleishaker D, Wollenhaupt J. Frequency and Duration of Early Non-serious Adverse Events in Patients with Rheumatoid Arthritis and Psoriatic Arthritis Treated with Tofacitinib. Rheumatol Ther. 2022 Apr;9(2):411-433. doi: 10.1007/s40744-021-00405-w. Epub 2021 Dec 17. PMID 34921355
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Bergman M, Tundia N, Yang M, Orvis E, Clewell J, Bensimon A. Economic Benefit from Improvements in Quality of Life with Upadacitinib: Comparisons with Tofacitinib and Methotrexate in Patients with Rheumatoid Arthritis. Adv Ther. 2021 Dec;38(12):5649-5661. doi: 10.1007/s12325-021-01930-4. Epub 2021 Oct 12. PMID 34636000
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Strand V, Kaine J, Alten R, Wallenstein G, Diehl A, Shi H, Germino R, Murray CW. Associations between Patient Global Assessment scores and pain, physical function, and fatigue in rheumatoid arthritis: a post hoc analysis of data from phase 3 trials of tofacitinib. Arthritis Res Ther. 2020 Oct 15;22(1):243. doi: 10.1186/s13075-020-02324-7. PMID 33059710
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Kivitz AJ, Cohen S, Keystone E, van Vollenhoven RF, Haraoui B, Kaine J, Fan H, Connell CA, Bananis E, Takiya L, Fleischmann R. A pooled analysis of the safety of tofacitinib as monotherapy or in combination with background conventional synthetic disease-modifying antirheumatic drugs in a Phase 3 rheumatoid arthritis population. Semin Arthritis Rheum. 2018 Dec;48(3):406-415. doi: 10.1016/j.semarthrit.2018.07.006. Epub 2018 Jul 19. PMID 30177460
- [Derived] Hall S, Nash P, Rischmueller M, Bossingham D, Bird P, Cook N, Witcombe D, Soma K, Kwok K, Thirunavukkarasu K. Tofacitinib, an Oral Janus Kinase Inhibitor: Pooled Efficacy and Safety Analyses in an Australian Rheumatoid Arthritis Population. Rheumatol Ther. 2018 Dec;5(2):383-401. doi: 10.1007/s40744-018-0118-2. Epub 2018 Jun 11. PMID 29949132
- [Derived] van Vollenhoven RF, Lee EB, Fallon L, Zwillich SH, Wilkinson B, Chapman D, DeMasi R, Keystone E. Tofacitinib in Rheumatoid Arthritis: Lack of Early Change in Disease Activity and the Probability of Achieving Low Disease Activity at Month 6. Arthritis Care Res (Hoboken). 2019 Jan;71(1):71-79. doi: 10.1002/acr.23585. PMID 29696833
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Genovese MC, van Vollenhoven RF, Wilkinson B, Wang L, Zwillich SH, Gruben D, Biswas P, Riese R, Takiya L, Jones TV. Switching from adalimumab to tofacitinib in the treatment of patients with rheumatoid arthritis. Arthritis Res Ther. 2016 Jun 23;18:145. doi: 10.1186/s13075-016-1049-3. PMID 27334658
- [Derived] Charles-Schoeman C, Burmester G, Nash P, Zerbini CA, Soma K, Kwok K, Hendrikx T, Bananis E, Fleischmann R. Efficacy and safety of tofacitinib following inadequate response to conventional synthetic or biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2016 Jul;75(7):1293-301. doi: 10.1136/annrheumdis-2014-207178. Epub 2015 Aug 14. PMID 26275429
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] van Vollenhoven RF, Fleischmann R, Cohen S, Lee EB, Garcia Meijide JA, Wagner S, Forejtova S, Zwillich SH, Gruben D, Koncz T, Wallenstein GV, Krishnaswami S, Bradley JD, Wilkinson B; ORAL Standard Investigators. Tofacitinib or adalimumab versus placebo in rheumatoid arthritis. N Engl J Med. 2012 Aug 9;367(6):508-19. doi: 10.1056/NEJMoa1112072. PMID 22873531
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921064&StudyName=A%20Phase%203%20Study%20Comparing%202%20Doses%20Of%20CP-690%2C550%20And%20The%20Active%20Comparator%2C%20Humira%20%28adalimumab%29%20Vs.%20Placebo%20For%20Treatment%20Of%20Rh

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg: CP-690,550 5 milligram (mg) tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
- CP-690,550 10 mg: CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
- Placebo, Then CP-690,550 5 mg: Placebo matched to CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week, for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve a minimum improvement of at least 20 percent (%) reduction in both swollen and tender joint counts from baseline, received CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12. At Month 6, remaining participants advanced to CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
- Placebo, Then CP-690,550 10 mg: Placebo matched to CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week, for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve a minimum improvement of at least 20% reduction in both swollen and tender joint counts from baseline, received CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12. At Month 6, remaining participants advanced to CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
- Adalimumab: Adalimumab 40 mg injection subcutaneously once every other week along with placebo matched to CP-690,550 5 mg tablet orally twice daily up to Month 12.
Period: Overall Study
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Started | 204 | 201 | 56 | 52 | 204
Completed | 150 | 158 | 47 | 39 | 162
Not Completed | 54 | 43 | 9 | 13 | 42
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 24 | 24 | 2 | 5 | 22
Not completed — Lack of Efficacy | 6 | 7 | 3 | 3 | 6
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 0 | 1 | 1
Not completed — Other | 18 | 9 | 4 | 4 | 12

BASELINE CHARACTERISTICS:
Groups:
- CP-690,550 5 mg: CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
- Placebo, Then CP-690,550 5 mg: Placebo matched to CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week, for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve a minimum improvement of at least 20% reduction in both swollen and tender joint counts from baseline, received CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12. At Month 6, remaining participants advanced to CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab | Total
Number analyzed (Participants) | 204 | 201 | 56 | 52 | 204 | 717
Age Continuous [Mean (Standard Deviation); unit: years] | 53.0 (11.9) | 52.9 (11.8) | 55.5 (13.7) | 51.9 (13.7) | 52.5 (11.7) | 52.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 168 | 43 | 39 | 162 | 586
  Male | 30 | 33 | 13 | 13 | 42 | 131

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 6
Description: ACR20 response: greater than or equal to (>=) 20% improvement in tender joint count (TJC); >= 20% improvement in swollen joint count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP). For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 6 analysis.
Time Frame: Month 6
Population: Full analysis set: all randomized participants who received >=1 dose and had >=1 post-baseline and baseline measurement (change from baseline endpoint). N(number of participants analyzed)=participants evaluable for this measure. Missing values due to withdrawal advancement to active treatment before Month 6 were imputed by non-responder imputation.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo matched to CP-690,550 tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction from baseline in both swollen and tender joint counts, received CP-690,550 5 mg or 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12. At Month 6, remaining participants received CP-690,550 5 mg or 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 196 | 196 | 106 | 199
percentage of participants | 51.53 | 52.55 | 28.30 | 47.24
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation for the difference in binomial proportions was used to test the superiority of CP-690,550 10 mg to placebo and 2-sided 95% confidence interval (CI) was evaluated for the difference in percentages; Test type: Superiority or Other; p < 0.0001, Normal approximation — A step-down procedure was used to control for multiple comparisons. In order for the comparison to 5 mg to be statistically significant, the comparison to 10 mg had to be statistically significant; Percent difference = 24.24, 95% CI 2-sided [13.18 to 35.31]
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; Normal approximation for the difference in binomial proportions was used to test the superiority of CP-690,550 5 mg to placebo and 2-sided 95% CI was evaluated for the difference in percentages; Test type: Superiority or Other; p < 0.0001, Normal approximation — [p-value comment as in outcome 1, analysis 1]; Percent difference = 23.22, 95% CI 2-sided [12.16 to 34.29]
Statistical Analysis 3: Comparison: Placebo vs Adalimumab; Normal approximation for the difference in binomial proportions was used to test the superiority of adalimumab to placebo and 2-sided 95% CI was evaluated for the difference in percentages; Test type: Superiority or Other; p = 0.0007, Normal approximation — Statistical testing was done at 5% significance level (2-sided); Percent difference = 18.93, 95% CI 2-sided [7.90 to 29.96]

2. Primary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) at Month 3
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; common activities over past week. Each item scored on 4-point scale from 0-3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as sum of domain scores and divided by number of domains answered. Total possible score range 0-3: 0=least difficulty and 3=extreme difficulty. For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 3 analysis.
Time Frame: Baseline, Month 3
Population: Full analysis set (FAS): all randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline and baseline measurement (for change from baseline endpoint). n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 201 | 199 | 106 | 201
units on a scale
  Baseline (n=201, 199, 106, 201) | 1.50 (0.64) | 1.53 (0.63) | 1.42 (0.68) | 1.50 (0.59)
  Month 3 (n=188, 185, 98, 190) | -0.49 (0.59) | -0.59 (0.58) | -0.17 (0.56) | -0.45 (0.52)
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Least squares (LS) mean difference and corresponding 95% CI was calculated using a mixed-effect repeated measure model with treatment, visit and treatment-by-visit interaction as fixed effect and participant as random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — A step-down procedure was used to control for multiple comparisons. For the comparison of 10 mg to placebo to be statistically significant in this measure, the comparison of 10 mg to placebo in ACR20 had to be significant; LS mean difference = -0.38, 95% CI 2-sided [-0.50 to -0.25], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; LS mean difference and corresponding 95% CI was calculated using a mixed-effect repeated measure model with treatment, visit and treatment-by-visit interaction as fixed effect and participant as random effect; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Step-down procedure: For the comparison of 5 mg to placebo to be statistically significant in this measure, the comparison of 10 mg to placebo as well as the comparison of 5 mg to placebo in ACR20 had to be statistically significant; LS mean difference = -0.31, 95% CI 2-sided [-0.43 to -0.19]
Statistical Analysis 3: Comparison: Placebo vs Adalimumab; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Statistical testing was done at 5% significance level (2-sided); LS mean difference = -0.25, 95% CI 2-sided [-0.37 to -0.13]

3. Primary Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) Less Than 2.6 at Month 6
Description: DAS28-4 (ESR) calculated from SJC and TJC using 28-joint count, erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PtGA) of disease activity (transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) less than or equal to (<=) 3.2 implied low disease activity and > 3.2 to 5.1 implied moderate to high disease activity, and < 2.6 = remission. For comparison of CP-690,550 with placebo, placebo sequences were combined into single reporting group for Month 6 analysis.
Time Frame: Month 6
Population: FAS: all randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline and baseline measurement (for change from baseline endpoint). N=participants evaluable for this measure. Missing values due to withdrawal advancement to active treatment before Month 6 were imputed using non-responder imputation (NRI).
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 177 | 176 | 92 | 178
percentage of participants | 6.21 | 12.50 | 1.09 | 6.74
Statistical Analysis 1: Comparison: CP-690,550 10 mg vs Placebo; Normal approximation to the binomial distribution was used to test the superiority of CP-690,550 10 mg to placebo and two-sided 95% CI was evaluated for the difference in percentages; Test type: Superiority or Other; p < 0.0001, Normal approximation — A step-down procedure was used to control for multiple comparisons. For comparison of 10 mg to placebo to be statistically significant in this measure, comparison of 10 mg to placebo in HAQ-DI had to be significant; Percent difference = 11.41, 95% CI 2-sided [6.08 to 16.73]
Statistical Analysis 2: Comparison: CP-690,550 5 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0151, Normal approximation — Step-down procedure: For the comparison of 5 mg to placebo to be statistically significant in this measure, the comparison of 10 mg to placebo as well as comparison of 5 mg to placebo in HAQ-DI had to be statistically significant; Percent difference = 5.12, 95% CI 2-sided [0.98 to 9.26]
Statistical Analysis 3: Comparison: Placebo vs Adalimumab; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.0091, Normal approximation — Statistical testing was done at 5% significance level (2-sided); Percent difference = 5.65, 95% CI 2-sided [1.40 to 9.90]

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 1 and 3
Description: ACR20 response: >=20% improvement in TJC; >= 20% improvement in SJC; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Month 1, 3
Population: FAS: all randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline and baseline measurement (for change from baseline endpoint). N=participants evaluable for this measure. Missing values due to withdrawal advancement to active treatment before Month 6 were imputed using NRI.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 196 | 196 | 106 | 199
percentage of participants
  Month 1 | 41.24 | 45.92 | 16.04 | 37.88
  Month 3 | 60.71 | 58.67 | 26.42 | 56.28

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Month 9 and 12
Description: ACR20 response: >=20% improvement in tender joint count; >=20% improvement in swollen joint count; and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Month 9, 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Groups:
- Placebo, Then CP-690,550 10 mg: Placebo matched to CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week, for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve a minimum improvement of at least 20 percent (%) reduction in both swollen and tender joint counts from baseline, received CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12. At Month 6, remaining participants advanced to CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 196 | 196 | 56 | 50 | 199
percentage of participants
  Month 9 | 49.49 | 50.51 | 30.36 | 36.00 | 47.24
  Month 12 | 49.49 | 49.49 | 33.93 | 34.00 | 49.25

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Month 1, 3 and 6
Description: ACR50 response: >=50% improvement in tender joint count; >=50% improvement in swollen joint count; and 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Month 1, 3, 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 196 | 196 | 106 | 199
percentage of participants
  Month 1 | 14.95 | 16.33 | 4.72 | 12.12
  Month 3 | 34.18 | 27.55 | 6.60 | 23.62
  Month 6 | 36.73 | 34.69 | 12.26 | 27.64

7. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Month 9 and 12
Description: as for outcome 6
Time Frame: Month 9, 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 196 | 196 | 56 | 50 | 199
percentage of participants
  Month 9 | 35.71 | 37.24 | 17.86 | 26.00 | 29.15
  Month 12 | 36.73 | 35.71 | 21.43 | 28.00 | 33.67

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Month 1, 3 and 6
Description: ACR70 response: >=70% improvement in tender joint count; >=70% improvement in swollen joint count; and 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Month 1, 3, 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 196 | 196 | 106 | 199
percentage of participants
  Month 1 | 2.58 | 4.08 | 0.94 | 3.03
  Month 3 | 12.24 | 14.80 | 1.89 | 8.54
  Month 6 | 19.90 | 21.94 | 1.89 | 9.05

9. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Month 9 and 12
Description: as for outcome 8
Time Frame: Month 9, 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 196 | 196 | 56 | 50 | 199
percentage of participants
  Month 9 | 18.37 | 21.94 | 8.93 | 10.00 | 11.06
  Month 12 | 22.96 | 23.47 | 10.71 | 14.00 | 16.58

10. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Baseline, Month 1, 3 and 6
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (milligram per liter [mg/L]). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 1, 3, 6
Population: FAS: all randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline and baseline measurement (for change from baseline endpoint). N=participants evaluable for this measure. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 200 | 199 | 106 | 201
units on a scale
  Baseline (n=200, 199, 106, 201) | 5.43 (0.89) | 5.43 (0.83) | 5.44 (0.88) | 5.33 (0.92)
  Month 1 (n=193, 196, 104, 197) | 4.26 (1.09) | 4.21 (1.05) | 5.09 (1.15) | 4.27 (1.06)
  Month 3 (n=187, 184, 99, 190) | 3.78 (1.21) | 3.77 (1.21) | 4.83 (1.25) | 3.88 (1.15)
  Month 6 (n=174, 180, 46, 181) | 3.51 (1.27) | 3.29 (1.22) | 3.85 (1.14) | 3.63 (1.19)

11. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Month 9 and 12
Description: DAS28-3 (CRP) was calculated from SJC and TJC using 28 joint count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Month 9, 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 160 | 167 | 49 | 41 | 171
units on a scale
  Month 9 (n=160, 167, 49, 41, 171) | 3.13 (1.11) | 3.20 (1.20) | 3.11 (1.11) | 3.03 (1.10) | 3.46 (1.21)
  Month 12 (n=149, 150, 48, 37, 160) | 3.05 (1.13) | 3.00 (1.18) | 3.12 (0.96) | 3.02 (1.28) | 3.18 (1.25)

12. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Baseline, Month 1, 3 and 6
Description: DAS28-4 (ESR) calculated from SJC and TJC using 28 joint count, ESR (mm/hour) and PGA of disease activity (participant rated arthritis activity assessment with transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 195 | 194 | 103 | 194
units on a scale
  Baseline (n=195, 194, 103, 194) | 6.56 (0.93) | 6.48 (0.89) | 6.45 (0.90) | 6.36 (0.93)
  Month 1 (n=172, 175, 90, 176) | 5.23 (1.19) | 5.14 (1.26) | 5.93 (1.22) | 5.13 (1.21)
  Month 3 (n=170, 166, 87, 167) | 4.64 (1.33) | 4.66 (1.39) | 5.60 (1.31) | 4.66 (1.28)
  Month 6 (n=155, 162, 41, 158) | 4.40 (1.38) | 4.21 (1.38) | 4.61 (1.17) | 4.37 (1.30)

13. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Month 9 and 12
Description: as for outcome 12
Time Frame: Month 9, 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 140 | 151 | 45 | 35 | 149
units on a scale
  Month 9 (n=140, 151, 45, 35, 149) | 4.00 (1.21) | 4.08 (1.33) | 3.99 (1.25) | 3.93 (1.17) | 4.20 (1.39)
  Month 12 (n=134, 136, 44, 32, 139) | 3.85 (1.22) | 3.88 (1.35) | 4.00 (0.95) | 3.70 (1.24) | 3.95 (1.48)

14. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (4 Variables) (DAS28-4 [CRP])
Description: DAS28-4 [CRP] calculated from SJC and TJC using 28 joint count, CRP (mg/L) and PGA of disease activity (participant rated arthritis activity assessment with transformed score ranging 0 to 10; higher score indicated greater affectation due to disease activity). Total score range:0 to 9.4, higher score indicated more disease activity. DAS28-4 (CRP) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 1, 3, 6, 9, 12
Population: Data was not analyzed for DAS28-4 (CRP) due to change in planned analyses.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (3 Variables) (DAS28-3 [ESR])
Description: DAS28-3 (ESR) was calculated from SJC and TJC using 28 joint count and ESR (mm/hour). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (ESR) =<3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Baseline, Month 1, 3, 6, 9, 12
Population: Data was not analyzed for DAS28-3 (ESR) due to change in planned analyses.
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) at Month 1, 3 and 6
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; common activities over past week. Each item scored on 4-point scale from 0-3:0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as sum of domain scores and divided by number of domains answered. Total possible score range 0-3: 0=least difficulty and 3=extreme difficulty.
Time Frame: Month 1, 3, 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 194 | 196 | 106 | 198
units on a scale
  Month 1 (n=194, 196, 106, 198) | 1.15 (0.66) | 1.11 (0.67) | 1.32 (0.69) | 1.12 (0.64)
  Month 3 (n=188, 185, 99, 190) | 1.00 (0.72) | 0.94 (0.75) | 1.25 (0.67) | 1.05 (0.64)
  Month 6 (n=174, 181, 46, 180) | 0.92 (0.72) | 0.89 (0.69) | 1.15 (0.71) | 0.98 (0.65)

17. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) at Month 9 and 12
Description: as for outcome 16
Time Frame: Month 9, 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 158 | 167 | 49 | 41 | 171
units on a scale
  Month 9 (n=158, 167, 49, 41, 171) | 0.86 (0.66) | 0.85 (0.66) | 0.89 (0.69) | 0.90 (0.64) | 0.97 (0.67)
  Month 12 (n=149, 149, 49, 38, 159) | 0.83 (0.68) | 0.81 (0.71) | 0.88 (0.71) | 0.91 (0.72) | 0.90 (0.67)

18. Secondary Outcome: Patient Assessment of Arthritis Pain at Baseline, Month 1, 3 and 6
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) visual analogue scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Month 1, 3, 6
Population: FAS: all randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline and baseline measurement (for change from baseline endpoint). n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 201 | 199 | 106 | 201
mm
  Baseline (n=201, 199, 106, 201) | 59.29 (20.95) | 59.01 (22.18) | 55.20 (21.27) | 56.46 (21.92)
  Month 1 (n=194, 196, 106, 198) | 39.71 (22.60) | 36.77 (22.63) | 49.92 (23.94) | 39.27 (24.29)
  Month 3 (n=188, 185, 99, 190) | 32.98 (23.09) | 31.27 (22.39) | 48.53 (23.42) | 36.27 (25.67)
  Month 6 (n=174, 181, 46, 179) | 30.40 (23.26) | 28.36 (22.52) | 35.04 (20.95) | 32.78 (22.57)

19. Secondary Outcome: Patient Assessment of Arthritis Pain at Month 9 and 12
Description: Participants rated the severity of arthritis pain on a 0 to 100 mm VAS, where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Month 9, 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 158 | 167 | 49 | 41 | 171
mm
  Month 9 (n=158, 167, 49, 41, 171) | 27.04 (21.35) | 27.99 (22.97) | 31.31 (22.66) | 24.93 (19.38) | 32.70 (24.18)
  Month 12 (n=150, 150, 49, 38, 160) | 26.99 (21.97) | 24.55 (20.68) | 28.23 (17.86) | 29.37 (20.57) | 27.94 (22.70)

20. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Baseline, Month 1, 3 and 6
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm VAS, where 0 mm = very well and 100 mm = very poorly.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 201 | 199 | 106 | 201
mm
  Baseline (n=201, 199, 106, 201) | 59.86 (21.38) | 56.55 (23.83) | 54.46 (21.27) | 57.22 (22.22)
  Month 1 (n=194, 196, 105, 197) | 41.85 (23.02) | 36.61 (23.51) | 50.70 (24.24) | 39.32 (23.83)
  Month 3 (n=188, 185, 99, 190) | 35.56 (23.81) | 31.25 (22.23) | 49.84 (22.45) | 36.97 (25.28)
  Month 6 (n=174, 181, 46, 180) | 32.79 (25.56) | 29.74 (22.41) | 37.76 (20.86) | 33.50 (21.97)

21. Secondary Outcome: Patient Global Assessment (PtGA) of Arthritis Pain at Month 9 and 12
Description: as for outcome 20
Time Frame: Month 9, 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 158 | 167 | 49 | 41 | 171
mm
  Month 9 (n=158, 167, 49, 41, 171) | 28.39 (22.31) | 29.47 (21.99) | 31.78 (20.75) | 30.00 (20.31) | 34.38 (24.93)
  Month 12 (n=149, 150, 49, 37, 160) | 26.86 (22.44) | 27.70 (22.09) | 30.78 (17.65) | 29.70 (20.69) | 30.33 (24.46)

22. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis Pain at Baseline, Month 1, 3 and 6
Description: Physician global assessment of arthritis was measured on a 0 to 100 mm VAS, where 0 mm = very good and 100 mm = very bad.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 199 | 199 | 106 | 201
mm
  Baseline (n=199, 199, 106, 201) | 59.92 (16.77) | 59.56 (16.70) | 60.28 (16.55) | 58.64 (15.98)
  Month 1 (n=193, 195, 106, 197) | 38.90 (18.56) | 36.16 (19.27) | 50.73 (22.08) | 38.81 (20.08)
  Month 3 (n=186, 185, 99, 189) | 30.28 (20.71) | 29.91 (21.04) | 45.12 (22.77) | 32.40 (21.08)
  Month 6 (n=174, 180, 46, 178) | 24.97 (19.26) | 24.46 (19.78) | 29.76 (20.43) | 27.77 (18.36)

23. Secondary Outcome: Physician Global Assessment (PGA) of Arthritis Pain at Month 9 and 12
Description: as for outcome 22
Time Frame: Month 9, 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 160 | 167 | 49 | 41 | 170
mm
  Month 9 (n=160, 167, 49, 41, 170) | 19.93 (16.20) | 21.92 (17.87) | 25.82 (20.32) | 23.78 (15.54) | 25.45 (19.94)
  Month 12 (n=149, 150, 48, 38, 157) | 18.67 (16.18) | 18.87 (16.05) | 19.77 (13.88) | 20.68 (14.51) | 20.44 (16.94)

24. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Baseline, Month 1, 3 and 6
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) and was reported as 2 summary scores; Physical Component Score and Mental Component Score. Total score range for the summary scores = 0-100 where higher scores represented higher level of functioning.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 201 | 199 | 106 | 201
units on a scale
  Baseline: Physical functioning (n=201,199,106,201) | 32.02 (9.48) | 31.06 (9.52) | 32.23 (9.43) | 31.74 (8.95)
  Baseline: Role physical (n=201,199,106,201) | 34.00 (9.11) | 33.54 (9.12) | 34.70 (8.01) | 34.79 (8.69)
  Baseline: Social functioning (n=201,199,106,201) | 36.15 (10.76) | 36.27 (11.59) | 39.36 (11.17) | 36.23 (11.52)
  Baseline: Bodily pain (n=201,199,106,201) | 33.42 (7.51) | 33.29 (7.42) | 34.53 (6.57) | 33.14 (7.33)
  Baseline: Mental health (n=201,199,106,201) | 39.04 (11.42) | 39.15 (11.19) | 41.11 (10.51) | 39.64 (11.19)
  Baseline: Role emotional (n=201,199,106,201) | 34.15 (12.49) | 34.11 (12.63) | 37.32 (11.97) | 35.54 (12.05)
  Baseline: Vitality (n=201,199,106,201) | 40.62 (9.23) | 40.79 (9.36) | 42.67 (8.85) | 39.95 (9.54)
  Baseline: General health (n=201,199,106,201) | 35.22 (8.95) | 35.81 (8.93) | 36.29 (8.38) | 35.18 (7.96)
  Baseline:Mental component (n=201,199,106,201) | 39.82 (11.68) | 40.21 (11.14) | 43.29 (10.58) | 40.58 (11.64)
  Baseline: Physical component (n=201,199,106,201) | 33.10 (7.69) | 32.62 (7.78) | 33.02 (6.23) | 32.74 (6.83)
  Month 1: Physical functioning (n=194,196,106,198) | 35.29 (9.94) | 35.23 (10.57) | 34.00 (9.68) | 35.38 (9.79)
  Month 1: Role physical (n=194,196,106,198) | 38.19 (9.34) | 38.45 (10.01) | 36.79 (9.39) | 38.37 (9.06)
  Month 1: Social functioning (n=194,196,106,198) | 40.77 (10.53) | 42.22 (10.64) | 41.74 (10.72) | 40.98 (10.41)
  Month 1: Bodily pain (n=194,196,106,198) | 40.14 (8.54) | 40.73 (8.46) | 36.18 (7.52) | 39.58 (8.36)
  Month 1: Mental health (n=194,196,106,198) | 42.31 (10.30) | 43.35 (11.13) | 41.79 (10.91) | 42.83 (10.93)
  Month 1: Role emotional (n=194,196,106,198) | 38.29 (12.54) | 38.64 (12.05) | 38.18 (11.89) | 39.10 (11.55)
  Month 1: Vitality (n=194,196,106,198) | 45.24 (9.33) | 46.99 (9.58) | 43.71 (8.74) | 44.44 (10.00)
  Month 1: General health (n=194,196,106,198) | 38.53 (9.24) | 39.98 (9.16) | 37.41 (8.61) | 38.35 (8.43)
  Month 1: Mental component (n=194,196,106,198) | 43.56 (10.60) | 44.92 (11.21) | 44.03 (11.04) | 44.05 (10.79)
  Month 1: Physical component (n=194,196,106,198) | 37.50 (7.99) | 37.86 (8.11) | 35.01 (7.36) | 37.08 (7.88)
  Month 3: Physical functioning (n=187,185,99,190) | 38.11 (10.39) | 38.49 (11.12) | 34.77 (8.92) | 36.56 (10.24)
  Month 3: Role physical (n=188,185,99,190) | 39.79 (9.55) | 40.93 (10.40) | 37.25 (8.88) | 39.51 (8.89)
  Month 3: Social functioning (n=188,185,99,190) | 41.59 (11.04) | 44.34 (11.00) | 41.41 (10.08) | 40.84 (10.92)
  Month 3: Bodily pain (n=187,185,99,190) | 41.08 (9.15) | 43.09 (9.58) | 37.05 (7.91) | 40.60 (9.54)
  Month 3: Mental health (n=188,185,99,190) | 42.43 (11.02) | 44.79 (11.25) | 42.44 (10.04) | 43.05 (10.45)
  Month 3: Role emotional (n=188,185,99,190) | 38.74 (12.56) | 41.76 (12.66) | 38.59 (12.42) | 39.24 (11.53)
  Month 3: Vitality (n=188,185,99,190) | 45.63 (9.91) | 48.09 (10.79) | 44.06 (9.22) | 45.57 (9.76)
  Month 3: General health (n=188,185,99,189) | 39.15 (9.52) | 41.35 (8.93) | 37.51 (8.08) | 39.33 (9.32)
  Month 3: Mental component (n=187,185,99,189) | 43.31 (11.47) | 46.49 (11.45) | 44.20 (10.65) | 43.90 (10.84)
  Month 3: Physical component (n=187,185,99,189) | 39.57 (8.76) | 40.30 (8.94) | 35.59 (7.33) | 38.58 (8.36)
  Month 6: Physical functioning (n=173,181,46,179) | 39.31 (10.92) | 38.56 (11.35) | 37.00 (8.99) | 37.29 (10.40)
  Month 6: Role physical (n=173,181,46,179) | 40.42 (10.03) | 41.29 (9.73) | 38.62 (7.95) | 39.99 (9.14)
  Month 6: Social functioning (n=173,181,46,180) | 43.85 (11.17) | 43.98 (11.30) | 42.49 (9.92) | 42.36 (10.43)
  Month 6: Bodily pain (n=173,181,46,180) | 42.79 (9.41) | 43.63 (9.31) | 39.79 (8.05) | 41.59 (8.95)
  Month 6: Mental health (n=173,181,46,180) | 44.31 (11.29) | 45.32 (11.43) | 41.21 (11.70) | 43.13 (11.35)
  Month 6: Role emotional (n=173,181, 46,179) | 40.78 (12.03) | 40.68 (11.77) | 39.22 (11.82) | 39.54 (11.85)
  Month 6: Vitality (n=173,181,46,180) | 47.35 (10.37) | 48.66 (10.08) | 45.06 (9.36) | 45.93 (9.88)
  Month 6: General health (n=173,180,46,180) | 40.53 (9.44) | 41.95 (8.89) | 39.03 (9.30) | 39.91 (8.72)
  Month 6: Mental component (n=173,180,46,179) | 45.44 (11.19) | 46.14 (11.43) | 43.43 (10.60) | 44.24 (11.69)
  Month 6: Physical component (n=173,180,46,179) | 40.45 (9.29) | 40.86 (8.71) | 38.44 (6.67) | 39.36 (8.39)

25. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) at Month 9 and 12
Description: as for outcome 24
Time Frame: Month 9, 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 159 | 167 | 49 | 41 | 171
units on a scale
  Month 9: Physical functioning(n=158,167,49,41,171) | 39.77 (10.29) | 38.74 (11.31) | 38.94 (9.81) | 38.59 (10.08) | 38.75 (10.23)
  Month 9: Role physical (n=159,167,49,41,171) | 41.66 (9.62) | 40.55 (10.15) | 41.77 (8.36) | 39.75 (9.20) | 41.12 (9.44)
  Month 9: Social functioning (n=159,167,49,41,171) | 43.52 (10.65) | 44.42 (9.96) | 44.55 (9.82) | 42.76 (9.78) | 42.03 (11.55)
  Month 9: Bodily pain (n=159,166,49,41,171) | 43.45 (9.02) | 42.75 (9.50) | 44.68 (8.86) | 42.26 (7.77) | 41.81 (9.73)
  Month 9: Mental health (n=159,166,49,41,171) | 44.47 (10.27) | 45.42 (10.44) | 44.83 (10.70) | 43.70 (10.16) | 43.44 (12.04)
  Month 9: Role emotional (n=159,167,49,41,171) | 39.98 (11.99) | 40.58 (12.07) | 39.84 (11.40) | 41.46 (11.81) | 40.07 (12.15)
  Month 9: Vitality (n=159,166,49,41,171) | 47.76 (9.51) | 48.69 (9.68) | 47.80 (8.94) | 46.41 (10.03) | 46.11 (10.28)
  Month 9: General health (n=159,166,49,41,171) | 41.15 (9.79) | 41.34 (9.20) | 41.39 (8.54) | 40.57 (9.34) | 40.12 (9.58)
  Month9:Mental component (n=158,165,49,41,171) | 44.79 (10.76) | 46.55 (10.52) | 45.31 (9.75) | 45.23 (11.22) | 44.08 (11.45)
  Month 9: Physical component (n=158,165,49,41,171) | 41.55 (8.57) | 40.32 (9.44) | 41.65 (8.20) | 39.73 (7.73) | 40.35 (8.31)
  Month 12:Physical functioning(n=149,149,49,38,160) | 40.16 (10.25) | 40.34 (11.59) | 39.24 (10.07) | 40.42 (9.84) | 39.21 (10.63)
  Month 12: Role physical (n=150,150,49,38,160) | 41.15 (9.35) | 42.34 (10.32) | 40.16 (8.73) | 41.18 (9.30) | 41.07 (9.29)
  Month 12: Social functioning (n=150,150,49,38,160) | 43.14 (10.46) | 44.07 (10.44) | 43.78 (9.97) | 44.94 (9.78) | 42.96 (10.92)
  Month 12: Bodily pain (n=150,150,49,38,160) | 43.44 (9.48) | 44.02 (10.02) | 43.90 (8.28) | 43.18 (7.76) | 42.73 (9.77)
  Month 12: Mental health (n=150,149,49,38,159) | 44.83 (10.02) | 45.06 (10.49) | 44.09 (9.20) | 45.28 (10.94) | 44.23 (10.93)
  Month 12:Role emotional (n=150,150,49,38,159) | 40.18 (11.46) | 42.25 (11.68) | 40.23 (10.79) | 41.03 (12.67) | 39.89 (11.63)
  Month 12: Vitality (n=150,149,49,38,159) | 47.60 (9.01) | 49.12 (9.95) | 47.31 (9.13) | 48.17 (9.36) | 46.27 (9.65)
  Month 12:General health (n=150,150,49,38,160) | 41.07 (9.85) | 42.33 (9.05) | 40.47 (9.44) | 40.77 (8.31) | 40.40 (9.13)
  Month 12:Mental component (n=149,149,49,38,158) | 45.02 (10.14) | 46.29 (10.56) | 45.02 (9.29) | 46.12 (11.75) | 44.42 (10.70)
  Month 12: Physical component(n=149,149,49,38,158) | 41.44 (8.81) | 41.96 (9.40) | 40.82 (8.01) | 41.12 (6.49) | 40.72 (8.84)

26. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT)-Fatigue Scale at Baseline, Month 1, 3 and 6
Description: FACIT-Fatigue scale is a 13-item questionnaire. Participant scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as 4 minus the participant's response. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflected an improvement in the participant's health status.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 201 | 199 | 106 | 201
units on a scale
  Baseline (n=201, 199, 106, 201) | 28.18 (10.48) | 28.56 (10.84) | 30.49 (10.23) | 27.95 (10.07)
  Month 1 (n=192, 196, 106, 198) | 32.54 (9.94) | 33.95 (10.54) | 31.66 (10.09) | 31.94 (10.48)
  Month 3 (n=187, 185, 99, 190) | 33.86 (10.18) | 35.12 (11.07) | 30.96 (10.21) | 32.72 (10.27)
  Month 6 (n=173, 181, 46, 180) | 34.58 (10.53) | 36.09 (10.07) | 32.37 (8.92) | 33.69 (10.58)

27. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT)-Fatigue Scale at Month 12
Description: as for outcome 26
Time Frame: Month 12
Population: FAS: all randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline and baseline measurement (for change from baseline endpoint). N=participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 150 | 151 | 49 | 38 | 159
units on a scale | 35.76 (9.53) | 37.53 (10.41) | 36.71 (7.81) | 35.71 (9.65) | 34.30 (9.83)

28. Secondary Outcome: Medical Outcomes Study-Sleep Scale (MOS-SS) at Baseline, Month 1, 3 and 6
Description: Participant-rated questionnaire to assess key constructs of sleep over the past week. Consists of a 12-item based on 7 sub scales: sleep disturbance (SD), snoring (Sno), awakened short of breath (ASOB) or with headache, sleep adequacy (Ade), and somnolence (Som) (range:0-100); sleep quantity (Qua)(range:0-24), and optimal (Opt) sleep (yes: 1, no: 0) and nine item index measures of sleep disturbance were constructed to provide composite scores: sleep problem summary (SPS) and overall sleep problems (OSP). Except sleep adequacy, optimal sleep and quantity, higher scores=greater impairment. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range* 100); total score range: 0 to 100; higher score = greater intensity of attribute.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 199 | 198 | 105 | 200
units on a scale
  Baseline: SPS (n=199, 198, 105, 200) | 42.13 (20.58) | 40.20 (19.48) | 39.14 (19.04) | 40.90 (19.68)
  Baseline: OSP (n=199, 198, 105, 200) | 43.24 (19.91) | 42.27 (19.32) | 41.27 (19.47) | 43.12 (19.50)
  Baseline: Ade (n=200, 198, 105, 200) | 42.95 (27.92) | 44.04 (28.21) | 47.43 (26.06) | 44.25 (27.83)
  Baseline: ASOB (n=200, 198, 105, 200) | 19.10 (24.91) | 15.96 (21.70) | 18.67 (24.54) | 20.00 (24.31)
  Baseline: SD (n=200, 198, 105, 200) | 45.46 (26.30) | 44.67 (25.96) | 43.95 (27.40) | 46.55 (26.31)
  Baseline: Qua (n=200, 198, 104, 199) | 6.46 (1.36) | 6.61 (1.70) | 6.70 (1.51) | 6.65 (1.82)
  Baseline: Sno (n=198, 197, 105, 199) | 36.06 (31.78) | 34.62 (31.71) | 30.10 (28.16) | 34.77 (30.50)
  Baseline: Som (n=199, 198, 105, 199) | 36.52 (21.22) | 35.66 (22.28) | 36.70 (20.55) | 33.47 (19.68)
  Month 1: SPS (n=194, 195, 105, 198) | 36.25 (19.19) | 34.03 (18.74) | 37.62 (18.83) | 38.16 (20.30)
  Month 1: OSP (n=194, 195, 105, 198) | 36.70 (18.13) | 34.81 (18.64) | 38.77 (18.45) | 39.18 (19.67)
  Month 1: Ade (n=194, 195, 105, 198) | 48.97 (27.11) | 52.62 (27.62) | 49.81 (25.87) | 46.87 (27.30)
  Month 1: ASOB (n=194, 195, 105, 198) | 18.35 (22.52) | 14.56 (20.13) | 19.81 (23.78) | 18.69 (25.26)
  Month 1: SD (n=194, 195, 105, 198) | 36.52 (23.48) | 35.46 (24.25) | 40.43 (26.13) | 39.41 (25.42)
  Month 1: Qua (n=193, 195, 105, 197) | 6.70 (1.38) | 6.97 (1.49) | 6.74 (1.49) | 6.89 (1.55)
  Month 1: Sno (n=194, 193, 104, 196) | 36.08 (32.53) | 34.30 (29.56) | 31.35 (27.13) | 32.76 (28.19)
  Month 1: Som (n=194, 195, 105, 198) | 31.68 (21.26) | 31.04 (22.02) | 33.90 (21.80) | 33.91 (19.60)
  Month 3: SPS (n=186, 185, 99, 190) | 35.39 (18.66) | 32.86 (20.91) | 37.54 (19.18) | 37.21 (20.47)
  Month 3: OSP (n=186, 185, 99, 190) | 35.74 (18.30) | 33.44 (20.23) | 38.55 (18.97) | 38.32 (20.05)
  Month 3: Ade (n=187, 185, 99, 190) | 50.59 (27.67) | 53.24 (28.90) | 48.99 (28.16) | 49.21 (28.65)
  Month 3: ASOB (n=187, 185, 99, 190) | 18.18 (22.12) | 14.81 (20.62) | 18.59 (20.85) | 18.42 (24.42)
  Month 3: SD (n=186, 185, 99, 190) | 35.93 (24.29) | 32.86 (25.10) | 38.66 (26.24) | 39.95 (25.83)
  Month 3: Qua (n=188, 185, 99, 190) | 6.82 (1.32) | 7.03 (1.45) | 6.51 (1.56) | 6.83 (1.47)
  Month 3: Sno (n=186, 184, 99, 189) | 33.66 (30.78) | 34.35 (30.06) | 30.10 (22.92) | 34.60 (27.80)
  Month 3: Som (n=187, 185, 99, 190) | 29.41 (19.66) | 30.74 (22.65) | 36.50 (20.10) | 31.05 (20.26)
  Month 6: SPS (n=173, 181, 46, 179) | 32.66 (18.60) | 31.79 (18.64) | 36.52 (19.89) | 36.31 (19.25)
  Month 6: OSP (n=173, 181, 46, 179) | 33.28 (17.93) | 32.46 (18.50) | 36.87 (18.51) | 36.73 (19.04)
  Month 6: Ade (n=173, 181, 46, 179) | 53.12 (28.85) | 53.76 (27.87) | 50.00 (26.83) | 50.22 (27.33)
  Month 6: ASOB (n=173, 181, 46, 179) | 16.65 (22.00) | 13.48 (20.21) | 16.52 (20.79) | 19.22 (22.37)
  Month 6: SD (n=173, 181, 46, 179) | 32.95 (23.76) | 32.00 (24.30) | 37.31 (24.73) | 36.39 (24.20)
  Month 6: Qua (n=173, 181, 45, 178) | 6.86 (1.18) | 7.10 (1.60) | 6.71 (1.50) | 6.81 (1.36)
  Month 6: Sno (n=171, 180, 46, 179) | 31.46 (31.43) | 35.00 (29.13) | 23.91 (23.33) | 33.18 (27.32)
  Month 6: Som (n=173, 181, 46, 179) | 28.17 (17.55) | 30.39 (22.37) | 33.62 (17.72) | 31.84 (20.38)

29. Secondary Outcome: Medical Outcomes Study-Sleep Scale (MOS-SS) at Month 12
Description: as for outcome 28
Time Frame: Month 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 148 | 150 | 49 | 37 | 158
units on a scale
  SPS (n=148, 150, 49, 37, 159) | 34.62 (18.58) | 30.64 (18.42) | 34.69 (19.10) | 34.68 (21.32) | 35.72 (20.25)
  OSP (n=148, 150, 49, 37, 158) | 34.86 (17.87) | 31.49 (17.90) | 36.00 (17.63) | 35.38 (20.40) | 36.52 (19.68)
  Ade (n=149, 150, 49, 37, 159) | 51.21 (26.96) | 57.20 (28.48) | 54.29 (27.84) | 50.00 (30.18) | 49.81 (27.20)
  ASOB (n=149, 150, 49, 37, 159) | 16.78 (19.74) | 14.13 (20.67) | 21.22 (22.14) | 18.38 (18.49) | 17.48 (21.79)
  SD (n=149, 150, 49, 37, 159) | 34.82 (23.95) | 32.32 (22.41) | 37.12 (23.55) | 34.86 (23.94) | 37.36 (25.19)
  Qua (n=148, 150, 49, 37, 158) | 6.78 (1.19) | 7.03 (1.47) | 6.86 (1.34) | 6.84 (1.34) | 6.72 (1.31)
  Sno (n=148, 150, 48, 37, 159) | 33.78 (29.95) | 30.53 (27.29) | 27.50 (22.83) | 32.43 (26.81) | 34.47 (30.01)
  Som (n=148, 150, 49, 37, 158) | 29.41 (18.95) | 27.07 (19.36) | 32.38 (17.53) | 29.37 (22.25) | 30.00 (21.21)

30. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study-Sleep Scale (MOS-SS) at Baseline, Month 1, 3 and 6
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence, sleep quantity and optimal sleep. Participants responded whether their sleep was optimal or not by choosing yes or no. Number of participants with optimal sleep are reported.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 201 | 199 | 106 | 201
participants
  Baseline (n=201, 199, 106, 201) | 94 | 94 | 49 | 88
  Month 1 (n=194, 196, 106, 198) | 93 | 107 | 55 | 95
  Month 3 (n=188, 185, 99, 190) | 100 | 110 | 37 | 93
  Month 6 (n=174, 181, 94, 182) | 100 | 100 | 46 | 93

31. Secondary Outcome: Number of Participants With Optimal Sleep Assessed Using Medical Outcomes Study-Sleep Scale (MOS-SS) at Month 12
Description: as for outcome 30
Time Frame: Month 12
Population: as for outcome 27
Measure: Number; unit: participants
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 150 | 151 | 49 | 38 | 160
participants | 80 | 84 | 28 | 19 | 75

32. Secondary Outcome: Euro Quality of Life-5 Dimension (EQ-5D) Health State Profile Utility Score at Baseline, Month 1, 3 and 6
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 200 | 199 | 106 | 201
units on a scale
  Baseline (n=200, 199, 106, 201) | 0.43 (0.32) | 0.43 (0.32) | 0.50 (0.28) | 0.45 (0.29)
  Month 1 (n=192, 195, 106, 198) | 0.61 (0.23) | 0.60 (0.25) | 0.56 (0.25) | 0.58 (0.27)
  Month 3 (n=187, 184, 99, 189) | 0.62 (0.28) | 0.64 (0.28) | 0.55 (0.27) | 0.61 (0.26)
  Month 6 (n=172, 180, 46, 178) | 0.66 (0.26) | 0.65 (0.25) | 0.58 (0.28) | 0.64 (0.24)

33. Secondary Outcome: Euro Quality of Life-5 Dimension (EQ-5D) Health State Profile Utility Score at Month 12
Description: as for outcome 32
Time Frame: Month 12
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 147 | 151 | 49 | 38 | 159
units on a scale | 0.69 (0.22) | 0.69 (0.22) | 0.68 (0.20) | 0.66 (0.19) | 0.66 (0.27)

34. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Month 3 and 6
Description: WLQ: participant-reported 25-item scale to evaluate degree to which health problems interfere with an ability to perform job roles along 4 dimensions: 5-items Time Management scale (TMS); 6-items Physical Demands scale (PDS); 9-items Mental-Interpersonal Demands Scale (MIDS); 5-items Output Demands scale (ODS). All the scales ranged from 0 (limited none of the time) to 100 (limited all of the time). Work Loss Index (WLI), which represented percentage of lost work over time period relative to a normative population, was derived (total score: 0 [no loss] to 100 [complete loss of work]).
Time Frame: Month 3, 6
Population: FAS: all randomized participants who received at least 1 dose of study drug, had at least 1 post-baseline and baseline measurement (for change from baseline endpoint). N=participants evaluable for this measure. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 85 | 81 | 42 | 78
units on a scale
  Baseline: TMS (n=79, 77, 40, 76) | 41.46 (23.42) | 42.09 (28.98) | 37.65 (23.69) | 46.43 (25.94)
  Baseline: PDS (n=85, 76, 40, 77) | 49.99 (23.16) | 52.14 (24.22) | 53.24 (23.62) | 44.51 (21.15)
  Baseline: MIDS (n=82, 79, 41, 77) | 26.80 (22.80) | 27.30 (22.32) | 24.85 (28.33) | 28.45 (23.77)
  Baseline: ODS (n=80, 74, 40, 77) | 36.34 (26.55) | 37.29 (28.16) | 29.28 (26.41) | 36.82 (22.71)
  Baseline: WLI (n=85, 81, 42, 81) | 9.76 (5.34) | 9.85 (5.67) | 8.83 (5.90) | 9.92 (5.01)
  Month 3: TMS (n=74, 68, 40, 70) | 31.31 (25.50) | 21.97 (25.52) | 34.26 (26.40) | 35.73 (28.50)
  Month 3: PDS (n=77, 72, 39, 76) | 53.03 (26.21) | 47.04 (33.97) | 55.57 (27.38) | 54.38 (28.15)
  Month 3: MIDS (n=78, 72, 41, 73) | 21.45 (22.03) | 15.14 (20.53) | 23.20 (26.04) | 22.64 (21.97)
  Month 3: ODS (n=75, 70, 39, 76) | 26.64 (23.61) | 19.31 (23.89) | 27.44 (25.18) | 26.57 (22.50)
  Month 3: WLI (n=80, 74, 41, 78) | 7.89 (5.12) | 5.92 (5.17) | 8.39 (5.73) | 8.23 (5.47)
  Month 6: PDS (n=66, 65, 15, 71) | 55.62 (30.05) | 53.57 (36.13) | 55.03 (29.84) | 52.17 (28.69)
  Month 6: TMS (n=68, 65, 16, 67) | 29.87 (26.81) | 21.30 (27.67) | 24.53 (24.19) | 29.70 (25.24)
  Month 6: MIDS (n=70, 68, 16, 71) | 17.50 (21.18) | 12.87 (22.77) | 18.26 (23.15) | 22.61 (22.38)
  Month 6: ODS (n=67, 67, 16, 69) | 23.18 (25.53) | 16.44 (23.79) | 19.69 (20.77) | 25.82 (22.93)
  Month 6: WLI (n= 70, 69, 16, 73) | 7.32 (5.47) | 5.69 (5.54) | 6.89 (4.90) | 7.84 (5.04)

35. Secondary Outcome: Work Limitations Questionnaire (WLQ) Score at Baseline and Month 12
Description: as for outcome 34
Time Frame: Baseline, Month 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 57 | 55 | 21 | 14 | 60
units on a scale
  TMS (n=55, 53, 20, 14, 57) | 25.59 (25.10) | 20.77 (28.68) | 32.69 (29.07) | 28.75 (28.26) | 26.57 (26.68)
  PDS (n=55, 52, 18, 14, 58) | 54.35 (32.96) | 55.69 (38.22) | 51.81 (32.57) | 59.02 (36.59) | 50.41 (33.98)
  MIDS (n=55, 51, 21, 14, 58) | 14.72 (19.96) | 13.96 (23.76) | 21.46 (27.11) | 19.44 (24.29) | 17.99 (20.10)
  ODS (n=57, 50, 19, 14, 58) | 20.51 (23.13) | 17.35 (27.77) | 27.11 (27.29) | 25.36 (29.64) | 21.55 (22.63)
  WLI (n=57, 55, 21, 14, 60) | 6.61 (5.07) | 5.78 (5.59) | 7.75 (6.53) | 8.06 (6.01) | 6.85 (5.21)

36. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Baseline, Month 3 and 6
Description: Rheumatoid Arthritis (RA)-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost: any RA/non-RA related medical/non-medical (NM) practitioner visit, nursing home, hospital, surgery, emergency room (ER) treatment, diagnostic tests, over-night stay, home healthcare (HC) services, aids/devices used. Indirect costs associated with functional disability: employment status, willingness to work, work disability due to RA, sick leave, part time work, ability to perform chores, chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale; higher score indicated higher medical cost.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 201 | 199 | 106 | 201
units on a scale
  Baseline: Seen any doctor (n=201, 199, 106, 201) | 1.16 (0.37) | 1.13 (0.34) | 1.15 (0.36) | 1.15 (0.36)
  Baseline: Treated in ER (n=201, 199, 106, 201) | 1.95 (0.23) | 1.93 (0.26) | 1.93 (0.25) | 1.94 (0.25)
  Baseline: Admitted overnight stay (n=11,14,6,12) | 0.45 (0.82) | 0.21 (0.43) | 0.17 (0.41) | 0.08 (0.29)
  Baseline: Hospitalization (n=201, 199, 106, 201) | 1.94 (0.24) | 1.97 (0.17) | 1.93 (0.25) | 1.95 (0.23)
  Baseline: Outpatient surgeries (n=200,199,106,201) | 1.96 (0.20) | 1.97 (0.17) | 1.98 (0.14) | 1.97 (0.18)
  Baseline: Diagnostic tests (n=200,199,106,200) | 1.81 (0.39) | 1.83 (0.37) | 1.82 (0.39) | 1.82 (0.39)
  Baseline: In nursing home (n=201, 199, 106, 201) | 1.99 (0.12) | 2.00 (0.00) | 2.00 (0.00) | 1.98 (0.14)
  Baseline: Home HC services (n=201, 198, 106, 201) | 1.99 (0.10) | 1.99 (0.10) | 1.99 (0.10) | 1.99 (0.12)
  Baseline:Required aids/devices (n=201,199,106,201) | 1.92 (0.28) | 1.86 (0.35) | 1.92 (0.28) | 1.91 (0.29)
  Baseline: Seen NM practitioner (n=201,199,106,201) | 1.99 (0.12) | 1.97 (0.17) | 1.98 (0.14) | 1.97 (0.17)
  Baseline: Currently employed (n=201,199,106,201) | 1.64 (0.48) | 1.65 (0.48) | 1.64 (0.48) | 1.65 (0.48)
  Baseline: Feel well enough to work (n=73,83,39,81) | 1.90 (0.30) | 1.89 (0.31) | 1.82 (0.39) | 1.80 (0.40)
  Baseline: Retired (n=80,88,45,89) | 1.41 (0.50) | 1.41 (0.49) | 1.40 (0.50) | 1.39 (0.49)
  Baseline: Lost job/retired early(n=66,82,39,81) | 1.50 (0.50) | 1.70 (0.46) | 1.74 (0.44) | 1.57 (0.50)
  Baseline: Unable to work due to RA (n=76,84,40,78) | 1.36 (0.48) | 1.37 (0.49) | 1.45 (0.50) | 1.37 (0.49)
  Baseline: Work disabled due to RA (n=66,82,40,79) | 1.56 (0.50) | 1.70 (0.46) | 1.70 (0.46) | 1.65 (0.48)
  Baseline: Sick leave due to RA (n=167,166,92,167) | 1.85 (0.36) | 1.86 (0.35) | 1.84 (0.37) | 1.83 (0.38)
  Baseline: Part time work (n=169,166,92,167) | 1.92 (0.27) | 1.92 (0.27) | 1.93 (0.25) | 1.94 (0.24)
  Baseline: Performed paid work(n=169,166,91,167) | 1.69 (0.46) | 1.70 (0.46) | 1.66 (0.48) | 1.67 (0.47)
  Baseline: Unable to do chores (n=201,199,105,198) | 1.41 (0.49) | 1.46 (0.50) | 1.53 (0.50) | 1.41 (0.49)
  Baseline: Chores by housekeeper(n=201,199,106,201) | 1.89 (0.32) | 1.90 (0.29) | 1.93 (0.25) | 1.91 (0.29)
  Baseline: Chores by family (n=200,199,106,201) | 1.50 (0.50) | 1.48 (0.50) | 1.62 (0.49) | 1.51 (0.50)
  Month 3: Seen any doctor (n=186,185,99,190) | 1.27 (0.45) | 1.28 (0.45) | 1.22 (0.42) | 1.29 (0.45)
  Month 3: Treated in ER (n=186,185,99,190) | 1.96 (0.20) | 1.96 (0.19) | 1.96 (0.20) | 1.95 (0.22)
  Month 3: Admitted overnight stay (n=8,8,4,9) | 0.25 (0.46) | 0.88 (0.99) | 0.00 (0.00) | 0.22 (0.44)
  Month 3: Hospitalization (n=185,185,99,190) | 1.98 (0.15) | 1.97 (0.16) | 1.99 (0.10) | 1.98 (0.12)
  Month 3: Outpatient surgeries (n=185,185,99,190) | 1.98 (0.13) | 1.98 (0.15) | 1.96 (0.20) | 1.97 (0.18)
  Month 3: Diagnostic tests (n=184,185,99,190) | 1.90 (0.30) | 1.87 (0.34) | 1.91 (0.29) | 1.89 (0.31)
  Month 3: In nursing home (n=185,185,99,190) | 1.99 (0.07) | 2.00 (0.00) | 2.00 (0.00) | 1.99 (0.10)
  Month 3: Home HC services (n=184,185,99,190) | 1.99 (0.07) | 2.00 (0.00) | 2.00 (0.00) | 2.00 (0.00)
  Month 3: Required aids/devices (n=185,185,99,190) | 1.94 (0.25) | 1.91 (0.29) | 1.92 (0.27) | 1.92 (0.28)
  Month 3: Seen NM practitioner (n=185,185,99,190) | 1.97 (0.16) | 2.00 (0.00) | 1.98 (0.14) | 1.98 (0.12)
  Month 3: Currently employed (n=185,185,99,190) | 1.62 (0.49) | 1.64 (0.48) | 1.63 (0.49) | 1.64 (0.48)
  Month 3: Feel well enough to work (n=74,79,41,80) | 1.70 (0.46) | 1.73 (0.44) | 1.93 (0.26) | 1.74 (0.44)
  Month 3: Retired (n=80,86,47,86) | 1.39 (0.49) | 1.34 (0.48) | 1.38 (0.49) | 1.38 (0.49)
  Month 3: Lost job/retired early(n=73,78,40,79) | 1.55 (0.50) | 1.59 (0.50) | 1.75 (0.44) | 1.65 (0.48)
  Month 3: Unable to work due to RA (n=76,83,44,77) | 1.42 (0.50) | 1.46 (0.50) | 1.45 (0.50) | 1.58 (0.50)
  Month 3: Work disabled due to RA (n=71,82,41,73) | 1.63 (0.49) | 1.68 (0.47) | 1.61 (0.49) | 1.74 (0.44)
  Month 3: Sick leave due to RA (n=153,146,85,157) | 1.93 (0.26) | 1.94 (0.24) | 1.81 (0.39) | 1.90 (0.29)
  Month 3: Part time work (n=153,145,85,155) | 1.95 (0.21) | 1.97 (0.16) | 1.94 (0.24) | 1.94 (0.25)
  Month 3: Performed paid work(n=153,145,85,157) | 1.73 (0.45) | 1.81 (0.39) | 1.68 (0.47) | 1.70 (0.46)
  Month 3: Unable to do chores(n=182,182,99,189) | 1.62 (0.49) | 1.71 (0.46) | 1.59 (0.50) | 1.66 (0.47)
  Month 3: Chores by housekeeper (n=184,183,99,190) | 1.91 (0.29) | 1.94 (0.24) | 1.93 (0.26) | 1.94 (0.24)
  Month 3: Chores by family (n=183,183,99,190) | 1.67 (0.47) | 1.74 (0.44) | 1.66 (0.48) | 1.68 (0.47)
  Month 6: Seen any doctor (n=173,180,45,179) | 1.25 (0.43) | 1.28 (0.45) | 1.27 (0.45) | 1.31 (0.46)
  Month 6: Treated in ER (n=173,180,46,179) | 1.93 (0.25) | 1.97 (0.18) | 1.91 (0.28) | 1.98 (0.15)
  Month 6: Admitted overnight stay (n=12,6,4,3) | 0.58 (0.67) | 0.17 (0.41) | 0.00 (0.00) | 0.00 (0.00)
  Month 6: Hospitalization (n=172,180,46,179) | 1.95 (0.22) | 1.97 (0.16) | 1.96 (0.21) | 1.99 (0.07)
  Month 6: Outpatient surgeries (n=173,180,46,178) | 1.98 (0.15) | 1.96 (0.19) | 1.98 (0.15) | 1.99 (0.11)
  Month 6: Diagnostic tests (n=173,180,46,178) | 1.87 (0.33) | 1.86 (0.35) | 1.89 (0.31) | 1.89 (0.31)
  Month 6: In nursing home (n=173,180,46,178) | 1.99 (0.11) | 2.00 (0.00) | 2.00 (0.00) | 2.00 (0.00)
  Month 6: Home HC services (n=173,180,46,177) | 1.99 (0.11) | 1.99 (0.11) | 2.00 (0.00) | 2.00 (0.00)
  Month 6: Required aids/devices (n=173,180,46,178) | 1.91 (0.28) | 1.91 (0.29) | 1.87 (0.34) | 1.92 (0.27)
  Month 6: Seen NM practitioner (n=173,180,45,178) | 2.00 (0.00) | 1.98 (0.13) | 2.00 (0.00) | 1.99 (0.07)
  Month 6: Currently employed (n=173,180,46,179) | 1.62 (0.49) | 1.66 (0.48) | 1.63 (0.49) | 1.63 (0.48)
  Month 6: Feel well enough to work (72,81,23,76) | 1.75 (0.44) | 1.77 (0.43) | 1.83 (0.39) | 1.71 (0.46)
  Month 6: Retired (n=77,87,22,82) | 1.32 (0.47) | 1.30 (0.46) | 1.32 (0.48) | 1.35 (0.48)
  Month 6: Lost job/retired early (n=70,82,22,72) | 1.57 (0.50) | 1.66 (0.48) | 1.68 (0.48) | 1.67 (0.47)
  Month 6: Unable to work due to RA (n=73,83,23,74) | 1.51 (0.50) | 1.54 (0.50) | 1.48 (0.51) | 1.57 (0.50)
  Month 6: Work disabled due to RA (n=67,80,22,72) | 1.72 (0.45) | 1.70 (0.46) | 1.73 (0.46) | 1.72 (0.45)
  Month 6: Sick leave due to RA (n=138,134,38,144) | 1.93 (0.25) | 1.93 (0.25) | 1.92 (0.27) | 1.94 (0.24)
  Month 6: Part time work (n=135,134,37,142) | 1.94 (0.24) | 1.96 (0.21) | 1.97 (0.16) | 1.95 (0.22)
  Month 6: Performed paid work (n=136,136,38,142) | 1.75 (0.43) | 1.80 (0.40) | 1.74 (0.45) | 1.76 (0.43)
  Month 6: Unable to do chores(n=171,178,45,175) | 1.70 (0.46) | 1.74 (0.44) | 1.62 (0.49) | 1.67 (0.47)
  Month 6: Chores by housekeeper (n=172,180,45,180) | 1.92 (0.27) | 1.94 (0.23) | 1.93 (0.25) | 1.96 (0.19)
  Month 6: Chores by family (n=172,180,46,180) | 1.72 (0.45) | 1.74 (0.44) | 1.67 (0.47) | 1.71 (0.45)

37. Secondary Outcome: Work Productivity and Healthcare Resource Utilization (HCRU) at Month 12
Description: RA-HCRU assessed healthcare usage during last 3 months for direct, indirect medical cost domains. Direct cost: visit to doctor, NM practitioner, nursing home, hospital, surgery, ER treatment, diagnostic tests, over-night stay, home HC services, and aids/devices used. Indirect costs associated with functional disability: employment status, willingness to work, work disability due to RA, sick leave, part time work, ability to perform chores, chores done by family/friends/housekeeper. Assessment was based on 0 to 2-point scale; higher score indicated higher medical cost.
Time Frame: Month 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 148 | 151 | 49 | 38 | 160
units on a scale
  Seen any doctor (n=148,151,49,38,160) | 1.31 (0.46) | 1.27 (0.45) | 1.24 (0.43) | 1.24 (0.43) | 1.23 (0.42)
  Treated in ER (n=149,151,49,38,160) | 1.98 (0.14) | 1.97 (0.18) | 2.00 (0.00) | 1.97 (0.16) | 1.96 (0.19)
  Admitted overnight stay (n=3,5,0,1,6) | 0.33 (0.58) | 0.20 (0.45) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.17 (0.41)
  Hospitalization (n=148,151,49,38,160) | 1.98 (0.14) | 1.97 (0.18) | 1.98 (0.14) | 1.97 (0.16) | 1.98 (0.14)
  Outpatient surgeries (n=148,151,49,38,160) | 1.97 (0.18) | 1.99 (0.11) | 2.00 (0.00) | 1.95 (0.23) | 1.97 (0.17)
  Diagnostic tests (n=149,151,49,38,159) | 1.94 (0.24) | 1.87 (0.33) | 1.88 (0.33) | 1.84 (0.37) | 1.86 (0.35)
  In nursing home (n=149,151,49,38,159) | 1.99 (0.12) | 2.00 (0.00) | 2.00 (0.00) | 2.00 (0.00) | 1.99 (0.08)
  Home HC services (n=148,151,49,38,159) | 2.00 (0.00) | 2.00 (0.00) | 2.00 (0.00) | 2.00 (0.00) | 1.99 (0.08)
  Required aids/devices (n=148,151,49,38,160) | 1.93 (0.26) | 1.92 (0.27) | 1.94 (0.24) | 1.92 (0.27) | 1.91 (0.29)
  Seen NM practitioner(n=149,151,49,38,160) | 1.98 (0.14) | 1.97 (0.16) | 1.98 (0.14) | 1.95 (0.23) | 2.00 (0.00)
  Currently employed (n=148,151,49,38,160) | 1.59 (0.49) | 1.68 (0.47) | 1.61 (0.49) | 1.61 (0.50) | 1.64 (0.48)
  Feel well enough to work (n=61,79,19,19,76) | 1.72 (0.45) | 1.75 (0.44) | 1.84 (0.37) | 1.84 (0.37) | 1.68 (0.47)
  Retired (n=64,84,21,19,80) | 1.25 (0.44) | 1.31 (0.47) | 1.19 (0.40) | 1.53 (0.51) | 1.35 (0.48)
  Lost job/retired early (n=58,75,19,18,75) | 1.53 (0.50) | 1.72 (0.45) | 1.68 (0.48) | 1.78 (0.43) | 1.67 (0.47)
  Unable to work due to RA (n=59,77,19,19,77) | 1.56 (0.50) | 1.61 (0.49) | 1.58 (0.51) | 1.58 (0.51) | 1.57 (0.50)
  Work disabled due to RA (n=58,76,19,18,75) | 1.64 (0.48) | 1.75 (0.44) | 1.79 (0.42) | 1.67 (0.49) | 1.67 (0.47)
  Sick leave due to RA (n=118,112,37,30,124) | 1.96 (0.20) | 1.96 (0.19) | 1.95 (0.23) | 2.00 (0.00) | 1.97 (0.18)
  Part time work (n=117,112,37,30,123) | 1.95 (0.22) | 1.99 (0.09) | 2.00 (0.00) | 2.00 (0.00) | 1.99 (0.09)
  Performed paid work (n=118,114,37,31,123) | 1.83 (0.38) | 1.82 (0.39) | 1.78 (0.42) | 1.71 (0.46) | 1.82 (0.38)
  Unable to do chores (n=146,150,47,38,154) | 1.81 (0.40) | 1.75 (0.44) | 1.79 (0.41) | 1.84 (0.37) | 1.73 (0.45)
  Chores by housekeeper (n=148,151,49,38,160) | 1.94 (0.24) | 1.97 (0.16) | 1.96 (0.20) | 1.95 (0.23) | 1.93 (0.25)
  Chores by family (n=145,151,49,38,160) | 1.76 (0.43) | 1.80 (0.40) | 1.84 (0.37) | 1.71 (0.46) | 1.71 (0.45)

38. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Baseline, Month 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA/non-RA related number of events including visits to doctor, non-medical practitioner, hospital ER treatment, hospitalizations, number of surgeries, diagnostic tests, and devices/aids used were reported.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 168 | 174 | 90 | 172
events
  Baseline: Doctor visits (n=168,174,90,172) | 4.26 (3.51) | 4.06 (3.57) | 4.50 (5.32) | 3.87 (3.74)
  Baseline: NM practitioners visits (n=3,6,2,6) | 1.33 (0.58) | 3.00 (1.79) | 4.50 (4.95) | 10.00 (10.51)
  Baseline: Hospital ER visits (n=12,14,7,12) | 1.08 (0.51) | 1.93 (1.59) | 1.57 (0.79) | 1.58 (1.73)
  Baseline: Number visits hospitalized(n=11,5,7,11) | 2.82 (5.71) | 1.00 (0.00) | 1.00 (0.00) | 1.27 (0.90)
  Baseline:Number of outpatient surgeries(n=8,6,2,7) | 1.13 (0.35) | 1.33 (0.82) | 1.00 (0.00) | 2.57 (4.16)
  Baseline:Non-study diagnostic tests(n=37,33,19,36) | 1.73 (1.04) | 1.79 (1.17) | 1.21 (0.54) | 1.64 (1.10)
  Baseline:RA related doctor visit(n=169,175,91,172) | 1.33 (1.03) | 1.17 (0.70) | 1.26 (0.81) | 1.19 (0.73)
  Baseline: RA related ER visit (n=11,14,6,12) | 0.64 (0.81) | 0.64 (0.74) | 0.17 (0.41) | 0.25 (0.45)
  Baseline: RA diagnostic tests (n=38,33,19,37) | 0.50 (0.76) | 0.55 (0.62) | 0.47 (0.61) | 0.84 (0.73)
  Baseline: RA related hospitalization (n=11,6,7,11) | 0.91 (0.83) | 0.67 (0.52) | 0.57 (0.79) | 0.82 (0.60)
  Baseline: RA related outpatient surgery(n=7,6,3,7) | 0.43 (0.79) | 0.33 (0.82) | 0.33 (0.58) | 0.43 (0.79)
  Baseline: RA related NM visit (n=3,6,2,6) | 0.67 (0.58) | 0.50 (0.84) | 1.00 (0.00) | 1.00 (0.63)
  Month 3: Doctor visits (n=136,138,78,136) | 3.62 (4.25) | 2.86 (2.99) | 3.27 (3.93) | 3.05 (2.87)
  Month 3: NM practitioners visits (n=5,0,2,2) | 2.40 (0.89) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 17.00 (21.21) | 7.50 (9.19)
  Month 3: Hospital ER visits (n=8,8,4,10) | 1.38 (0.74) | 1.00 (0.00) | 1.75 (1.50) | 1.90 (1.10)
  Month 3: Number visits hospitalized (n=4,6,1,3) | 1.50 (1.00) | 1.00 (0.00) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.00 (0.00)
  Month 3: Number of outpatient surgeries(n=3,4,4,6) | 1.67 (0.58) | 1.00 (0.00) | 1.00 (0.00) | 1.33 (0.52)
  Month 3: Non-study diagnostic tests (n=18,23,9,20) | 1.72 (1.41) | 1.52 (0.79) | 1.56 (0.88) | 1.45 (0.83)
  Month 3: RA related doctor visit(n=136,138,78,136) | 0.91 (0.75) | 0.92 (0.67) | 0.90 (0.71) | 0.93 (0.65)
  Month 3: RA related ER visit (n=8,8,4,9) | 0.25 (0.46) | 0.50 (0.76) | 0.00 (0.00) | 0.00 (0.00)
  Month 3: RA-diagnostic tests (n=19,24,9,21) | 0.11 (0.32) | 0.21 (0.51) | 0.11 (0.33) | 0.24 (0.44)
  Month 3: RA related hospitalization (n=4,6,1,3) | 0.00 (0.00) | 0.17 (0.41) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant were evaluable. | 0.67 (1.15)
  Month 3: RA related outpatient surgery (n=3,4,4,6) | 0.00 (0.00) | 0.25 (0.50) | 0.25 (0.50) | 0.00 (0.00)
  Month 3: RA related NM visit (n=5,0,2,2) | 0.60 (0.89) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 1.50 (0.71) | 0.50 (0.71)
  Month 6: Doctor visits (n=132,131,33,128) | 3.30 (4.17) | 2.86 (4.23) | 2.52 (1.91) | 2.73 (2.96)
  Month 6: NM practitioners visits (n=1,3,0,1) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 2.67 (2.89) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 14.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 6: Hospital ER visits (n=12,6,4,4) | 1.08 (0.29) | 1.17 (0.41) | 1.00 (0.00) | 1.75 (0.96)
  Month 6: Number visits hospitalized (n=9,5,2,1) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 6: Number of outpatient surgeries(n=4,7,1,2) | 1.25 (0.50) | 1.14 (0.38) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.50 (0.71)
  Month 6: Non-study diagnostic tests (n=21,25,5,19) | 2.33 (3.89) | 1.96 (1.31) | 1.80 (0.45) | 1.53 (0.61)
  Month 6: RA related doctor visit(n=132,131,33,129) | 0.81 (0.63) | 0.96 (0.74) | 0.88 (0.86) | 1.00 (0.56)
  Month 6: RA related ER visit (n=12,6,4,3) | 0.25 (0.62) | 0.67 (0.82) | 0.00 (0.00) | 0.00 (0.00)
  Month 6: RA-diagnostic tests (n=21,25,5,19) | 0.18 (0.50) | 0.16 (0.37) | 0.20 (0.45) | 0.11 (0.32)
  Month 6: RA related hospitalization (n=9,5,2,1) | 0.22 (0.67) | 0.40 (0.89) | 0.00 (0.00) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant were evaluable.
  Month 6: RA related outpatient surgery (n=4,7,1,2) | 0.00 (0.00) | 0.43 (0.79) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant were evaluable. | 1.00 (1.41)
  Month 6: RA related NM visit (n=1,3,0,1) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant were evaluable. | 0.67 (1.15) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable.

39. Secondary Outcome: Number of Events Including Visits, Surgeries, Tests or Devices as Assessed Using RA-HCRU at Month 12
Description: as for outcome 38
Time Frame: Month 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 104 | 111 | 37 | 30 | 125
events
  Doctor visit (n=102,111,37,30,125) | 2.73 (2.78) | 2.80 (2.46) | 3.92 (5.97) | 3.50 (3.34) | 2.94 (3.93)
  NM practitioners visits (n=3,4,1,2,0) | 10.67 (11.72) | 9.75 (10.97) | 192.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 10.50 (6.36) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point.
  Hospital ER visits (n=3,5,0,1,6) | 1.00 (0.00) | 2.40 (1.34) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 3.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.00 (0.00)
  Number of visits hospitalized (n=3,5,1,1,3) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.00 (0.00)
  Number of outpatient surgeries (n=5,2,0,2,5) | 1.40 (0.89) | 1.50 (0.71) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 1.00 (0.00) | 2.20 (2.17)
  Non-study diagnostic tests (n=8,19,6,6,22) | 1.13 (0.35) | 1.95 (1.31) | 3.17 (2.64) | 1.33 (0.82) | 1.64 (0.90)
  RA related doctor visit (n=104,111,37,30,125) | 0.82 (0.59) | 0.93 (0.57) | 0.89 (0.52) | 0.87 (0.68) | 0.84 (0.80)
  RA related ER visits (n=3,5,0,1,6) | 0.33 (0.58) | 0.00 (0.00) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.17 (0.41)
  RA-diagnostic tests (n=9,19,6,6,22) | 0.11 (0.33) | 0.21 (0.42) | 0.17 (0.41) | 0.00 (0.00) | 0.05 (0.21)
  RA related hospitalization (n=3,5,1,1,3) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (NA) — Standard deviation was not estimable since only 1 participant were evaluable. | 0.00 (NA) — Standard deviation was not estimable since only 1 participant were evaluable. | 0.67 (0.58)
  RA related outpatient surgery (n=5,2,0,2,5) | 0.00 (0.00) | 0.00 (0.00) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 0.00 (0.00) | 0.00 (0.00)
  RA related NM visits (n=3,4,1,2,0) | 0.00 (0.00) | 0.50 (1.00) | 0.00 (NA) — Standard deviation was not estimable as only 1 participant was evaluable. | 0.00 (0.00) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point.

40. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Baseline, Month 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of days spent in hospital, nursing home, aids/devices used, on sick leave, work per week, performed part time work, performed paid work, chores done by housekeeper and chores done by family/friends.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 101 | 102 | 39 | 97
days
  Baseline: Hospital length of stay (n=11,6,7,11) | 13.64 (12.91) | 10.83 (9.89) | 13.43 (9.78) | 12.82 (10.93)
  Baseline: Days in nursing home (n=3,0,0,4) | 19.33 (17.56) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 14.25 (9.95)
  Baseline: Days devices/aids used (n=17,28,8,16) | 133.88 (111.17) | 67.32 (61.88) | 172.75 (94.28) | 66.13 (65.33)
  Baseline: Days of work per week (n=71,69,38,70) | 4.94 (1.18) | 4.80 (1.05) | 4.95 (0.98) | 5.01 (1.04)
  Baseline: Chores by housekeeper (n=23,19,6,18) | 15.57 (25.73) | 14.95 (27.24) | 38.83 (41.44) | 6.94 (6.86)
  Baseline: Chores by family (n=101,102,39,97) | 24.06 (29.27) | 26.57 (31.02) | 26.95 (32.87) | 29.80 (32.91)
  Baseline: Days on sick leave (n=24,24,15,29) | 19.58 (27.78) | 16.33 (27.21) | 29.60 (34.88) | 16.31 (26.05)
  Baseline: Days of part time work (n=13,13,6,10) | 13.31 (18.94) | 25.31 (61.19) | 5.33 (3.44) | 18.50 (26.88)
  Baseline: Paid work, bothered by RA(n=51,47,31,53) | 29.10 (27.47) | 29.45 (31.37) | 28.74 (28.76) | 42.74 (31.81)
  Baseline: RA related devices/aids (n=17,28,9,17) | 1.76 (1.15) | 1.39 (0.69) | 2.33 (1.66) | 1.65 (1.06)
  Month 3: Hospital length of stay (n=4,6,1,3) | 6.25 (4.03) | 10.00 (10.75) | 2.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 10.33 (8.14)
  Month 3: Days in nursing home (n=0,0,0,2) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 17.50 (4.95)
  Month 3: Days devices/aids used (n=11,17,6,15) | 117.91 (112.91) | 60.41 (88.79) | 163.83 (153.63) | 91.80 (95.18)
  Month 3: Days of work per week (n=70,66,38,68) | 4.83 (0.95) | 4.68 (1.18) | 4.95 (0.80) | 4.75 (1.25)
  Month 3: Chores by housekeeper (n=17,11,7,12) | 12.59 (23.15) | 6.00 (8.63) | 8.00 (12.54) | 10.50 (16.08)
  Month 3: Chores by family (n=60,47,34,58) | 24.10 (32.38) | 18.32 (24.03) | 24.97 (31.72) | 25.41 (30.46)
  Month 3: Days on sick leave (n=11,9,17,15) | 24.27 (33.73) | 18.44 (29.37) | 27.12 (31.42) | 5.13 (4.60)
  Month 3: Days of part time work (n=7,4,6,10) | 13.29 (13.76) | 25.50 (27.77) | 5.50 (3.27) | 14.90 (27.04)
  Month 3: Paid work, bothered by RA (n=39,28,28,44) | 16.08 (21.77) | 26.57 (32.41) | 19.93 (20.79) | 33.61 (30.31)
  Month 3: RA related devices/aids (n=12,17,8,16) | 1.75 (1.22) | 1.12 (1.36) | 2.38 (1.60) | 1.81 (0.98)
  Month 6: Hospital length of stay (n=9,5,2,1) | 10.00 (8.20) | 12.80 (16.71) | 8.50 (2.12) | 6.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Month 6: Days in nursing home (n=2,0,0,0) | 27.00 (18.38) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point.
  Month 6: Days devices/aids used (n=14,16,5,14) | 102.29 (115.01) | 126.25 (134.08) | 80.20 (73.45) | 94.21 (76.92)
  Month 6: Days of work per week (n=65,61,17,66) | 4.94 (0.85) | 4.70 (1.09) | 5.35 (0.93) | 4.95 (0.92)
  Month 6: Chores by housekeeper (n=11,10,3,7) | 7.73 (8.25) | 15.80 (22.73) | 44.00 (42.57) | 7.29 (3.82)
  Month 6: Chores by family (n=46,46,15,50) | 13.59 (16.95) | 29.09 (35.16) | 35.53 (39.39) | 22.64 (29.51)
  Month 6: Days on sick leave (n=7,9,3,9) | 29.57 (41.48) | 12.44 (14.60) | 3.00 (2.00) | 8.67 (13.13)
  Month 6: Days of part time work (n=7,6,1,7) | 7.57 (6.80) | 24.67 (33.07) | 4.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 9.29 (8.67)
  Month 6: Paid work, bothered by RA (n=31,25,10,33) | 14.71 (18.47) | 20.40 (25.93) | 11.00 (9.13) | 24.55 (26.88)
  Month 6: RA related devices/aids (n=15,16,6,14) | 2.00 (1.73) | 1.56 (1.46) | 2.17 (1.83) | 2.07 (1.27)

41. Secondary Outcome: Number of Days as Assessed Using RA-HCRU at Month 12
Description: as for outcome 40
Time Frame: Month 12
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 60 | 49 | 19 | 15 | 58
days
  Hospital length of stay (n=3,5,1,1,3) | 8.00 (6.93) | 5.60 (2.70) | 15.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 15.33 (4.51)
  Days in nursing home (n=2,0,0,0,1) | 24.50 (4.95) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 10.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Days devices/aids used (n=11,12,3,2,15) | 144.55 (258.85) | 51.75 (41.51) | 163.67 (173.70) | 321.50 (327.39) | 79.33 (74.00)
  Days of work per week (n=60,49,19,15,58) | 4.83 (1.04) | 5.04 (0.93) | 5.16 (0.90) | 4.93 (0.70) | 4.95 (1.07)
  Chores by housekeeper (n=9,4,1,2,10) | 4.44 (3.40) | 7.75 (5.06) | 90.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 24.00 (16.97) | 4.90 (3.78)
  Chores by family (n=35,30,8,10,45) | 22.06 (27.84) | 13.13 (12.28) | 51.88 (40.91) | 28.40 (33.88) | 23.49 (28.68)
  Days on sick leave (n=5,3,2,0,4) | 10.40 (11.41) | 36.00 (45.97) | 50.00 (56.57) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 18.25 (14.06)
  Days of part time work (n=6,1,0,0,1) | 11.33 (12.55) | 33.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 30.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Paid work, bothered by RA (n=20,20,7,9,22) | 24.10 (30.75) | 20.40 (27.90) | 11.43 (8.60) | 12.33 (12.32) | 22.86 (24.20)
  RA related devices/aids used (n=11,12,3,3,15) | 2.18 (2.79) | 0.75 (0.62) | 2.33 (1.53) | 3.00 (2.65) | 1.53 (0.74)

42. Secondary Outcome: Number of Hours Per Day as Assessed RA-HCRU at Baseline, Month 3 and 6
Description: RA-HCRU assessed healthcare usage during previous 3 months for direct or indirect medical cost domains. Any RA or non-RA related number of hours spent per day for home healthcare services, chores done by housekeeper, chores done by family or friends, hours affected per day and average number of hours missed work per day were reported.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 101 | 102 | 39 | 95
hours per day
  Baseline: Home HC services (n=2,2,1,2) | 3.00 (2.83) | 1.50 (0.71) | 2.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 1.00 (0.00)
  Baseline: Work done (n=72,69,38,70) | 7.76 (2.40) | 7.54 (2.25) | 7.79 (1.76) | 8.16 (2.85)
  Baseline: Chores by housekeeper (n=22,19,7,18) | 5.23 (4.60) | 5.53 (5.36) | 8.00 (7.55) | 3.89 (2.37)
  Baseline: Chores by family (n=101,102,39,95) | 4.24 (4.75) | 3.31 (2.76) | 4.21 (4.71) | 2.82 (1.79)
  Baseline: Missed work due to RA (n=13,13,6,10) | 6.38 (7.22) | 5.00 (5.85) | 4.00 (1.26) | 4.00 (4.11)
  Baseline: RA related home HC services (n=2,2,1,3) | 0.50 (0.71) | 1.00 (0.00) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.33 (0.58)
  Month 3: Home HC services (n=1,0,0,0) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point.
  Month 3: Work done (n=70,66,38,68) | 8.06 (3.59) | 7.53 (1.92) | 8.53 (5.62) | 8.38 (4.89)
  Month 3: Chores by housekeeper (n=17,11,7,12) | 4.00 (2.12) | 5.73 (2.61) | 5.00 (2.00) | 4.17 (1.99)
  Month 3: Chores by family (n=59,46,34,59) | 3.46 (3.67) | 3.28 (2.60) | 3.41 (2.72) | 3.68 (3.72)
  Month 3: Missed work due to RA (n=7,4,6,9) | 4.57 (5.03) | 20.75 (39.51) | 5.50 (5.01) | 3.56 (1.59)
  Month 3: RA related home HC services (n=1,0,0,0) | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point.
  Month 6: Home HC services (n=2,2,0,0) | 2.50 (2.12) | 16.00 (5.66) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point.
  Month 6: Work done (n=65,61,17,66) | 8.35 (4.46) | 7.72 (2.24) | 9.71 (7.59) | 8.00 (4.27)
  Month 6: Chores by housekeeper (n=11,10,3,7) | 3.36 (2.58) | 5.40 (2.50) | 5.33 (1.53) | 6.29 (7.95)
  Month 6: Chores by family (n=47,45,13,51) | 3.30 (2.69) | 2.91 (2.00) | 3.69 (2.32) | 3.33 (3.55)
  Month 6: Missed work due to RA (n=7,6,1,7) | 4.57 (5.19) | 3.17 (2.32) | 5.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 3.29 (1.70)
  Month 6: RA related home HC services (n=2,2,0,0) | 1.00 (1.41) | 0.50 (0.71) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point.

43. Secondary Outcome: Number of Hours Per Day as Assessed RA-HCRU at Month 12
Description: as for outcome 42
Time Frame: Month 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 60 | 49 | 19 | 15 | 58
hours per day
  Home HC services (n=0,0,0,0,1) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Work done (n=60,49,19,15,58) | 7.52 (2.27) | 7.82 (1.60) | 9.53 (7.65) | 7.73 (2.40) | 7.93 (3.12)
  Chores by housekeeper (n=8,4,1,2,10) | 4.63 (3.16) | 4.75 (0.96) | 3.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 6.00 (1.41) | 4.10 (2.08)
  Chores by family (n=34,30,8,10,44) | 2.65 (1.95) | 4.00 (4.11) | 2.88 (2.17) | 2.70 (2.26) | 2.55 (1.81)
  Missed work due to RA (n=6,1,0,0,1) | 2.00 (1.67) | 4.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 4.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  RA related home HC services (n=0,0,0,0,1) | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | NA (NA) — Data not available as no participant was evaluable for the treatment arm at the given time point. | 1.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.

44. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Baseline, Month 3 and 6
Description: Work performance of participants on number of days bothered was based on 10-point scale, where higher score indicated lower work performance.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo | Adalimumab
Number analyzed (Participants) | 139 | 141 | 83 | 142
units on a scale
  Baseline (n=139,141,83,142) | 4.16 (3.05) | 4.16 (3.33) | 4.08 (3.32) | 4.19 (3.09)
  Month 3 (n=137,129,76,139) | 2.68 (2.75) | 2.81 (2.89) | 3.38 (2.84) | 3.09 (2.81)
  Month 6 (n=125,125,35,127) | 2.31 (2.51) | 2.39 (2.84) | 2.17 (2.64) | 2.66 (2.54)

45. Secondary Outcome: Work Performance in Past 3 Months on Days Bothered as Assessed Using RA-HCRU at Month 12
Description: as for outcome 44
Time Frame: Month 12
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 5 mg | CP-690,550 10 mg | Placebo, Then CP-690,550 5 mg | Placebo, Then CP-690,550 10 mg | Adalimumab
Number analyzed (Participants) | 101 | 101 | 32 | 30 | 107
units on a scale | 2.18 (2.65) | 1.92 (2.50) | 2.69 (2.66) | 2.23 (3.02) | 1.93 (2.45)

ADVERSE EVENTS:
Time Frame: Baseline Through Month 12
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- CP-690,550 5 mg (Up To Month 3): CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 3.
- CP-690,550 10 mg (Up To Month 3): CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 3.
- Placebo (Up To Month 3): Placebo matched to CP-690,550 tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week for 3 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction from baseline in both swollen and tender joint counts, received CP-690,550 5 mg or 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12. At Month 6, remaining participants received CP-690,550 5 mg or 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
- Adalimumab (Up To Month 3): Adalimumab 40 mg injection subcutaneously once every other week along with placebo matched to CP-690,550 5 mg tablet orally twice daily up to Month 3.
- CP-690,550 5 mg (Month 3 to 6): CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week from Month 3 to Month 6.
- CP-690,550 10 mg (Month 3 to 6): CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week from Month 3 to Month 6.
- Placebo (Month 3 to 6): Placebo matched to CP-690,550 tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week for 3 to 6 months. Response was assessed at Month 3 and participants who failed to achieve at least 20% reduction from baseline in both swollen and tender joint counts, received CP-690,550 5 mg or 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12. At Month 6, remaining participants received CP-690,550 5 mg or 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week up to Month 12.
- Adalimumab (Month 3 to 6): Adalimumab 40 mg injection subcutaneously once every other week along with placebo matched to CP-690,550 5 mg tablet orally twice daily from Month 3 to Month 6.
- CP-690,550 5 mg (Post Month 6): CP-690,550 5 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week from Month 6 to Month 12.
- CP-690,550 10 mg (Post Month 6): CP-690,550 10 mg tablet orally twice daily along with placebo matched to adalimumab 40 mg injection subcutaneously once every other week from Month 6 to Month 12.
- Adalimumab (Post Month 6): Adalimumab 40 mg injection subcutaneously once every other week along with placebo matched to CP-690,550 5 mg tablet orally twice daily from Month 6 to Month 12.
Arm/Group | CP-690,550 5 mg (Up To Month 3) | CP-690,550 10 mg (Up To Month 3) | Placebo (Up To Month 3) | Adalimumab (Up To Month 3) | CP-690,550 5 mg (Month 3 to 6) | CP-690,550 10 mg (Month 3 to 6) | Placebo (Month 3 to 6) | Adalimumab (Month 3 to 6) | CP-690,550 5 mg (Post Month 6) | CP-690,550 10 mg (Post Month 6) | Adalimumab (Post Month 6)
Serious Adverse Events (participants affected / at risk) | 12/204 | 10/201 | 2/108 | 5/204 | 10/232 | 7/222 | 2/59 | 6/204 | 11/260 | 10/253 | 7/204
Other Adverse Events (participants affected / at risk) | 51/204 | 44/201 | 18/108 | 50/204 | 18/232 | 8/222 | 3/59 | 18/204 | 36/260 | 44/253 | 24/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (Up To Month 3) (N=204) | CP-690,550 10 mg (Up To Month 3) (N=201) | Placebo (Up To Month 3) (N=108) | Adalimumab (Up To Month 3) (N=204) | CP-690,550 5 mg (Month 3 to 6) (N=232) | CP-690,550 10 mg (Month 3 to 6) (N=222) | Placebo (Month 3 to 6) (N=59) | Adalimumab (Month 3 to 6) (N=204) | CP-690,550 5 mg (Post Month 6) (N=260) | CP-690,550 10 mg (Post Month 6) (N=253) | Adalimumab (Post Month 6) (N=204)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gallbladder empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervix disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg (Up To Month 3) (N=204) | CP-690,550 10 mg (Up To Month 3) (N=201) | Placebo (Up To Month 3) (N=108) | Adalimumab (Up To Month 3) (N=204) | CP-690,550 5 mg (Month 3 to 6) (N=232) | CP-690,550 10 mg (Month 3 to 6) (N=222) | Placebo (Month 3 to 6) (N=59) | Adalimumab (Month 3 to 6) (N=204) | CP-690,550 5 mg (Post Month 6) (N=260) | CP-690,550 10 mg (Post Month 6) (N=253) | Adalimumab (Post Month 6) (N=204)
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 7 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 3 | 1 | 4 | 0 | 0 | 0 | 0 | 7 | 10 | 4
Herpes zoster (Infections and infestations) | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 4
Nasopharyngitis (Infections and infestations) | 8 | 4 | 0 | 7 | 5 | 2 | 1 | 3 | 8 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 9 | 7 | 1 | 7 | 0 | 0 | 0 | 0 | 9 | 6 | 4
Urinary tract infection (Infections and infestations) | 5 | 2 | 0 | 7 | 5 | 1 | 0 | 6 | 2 | 4 | 5
Alanine aminotransferase increased (Investigations) | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 5 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 7 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 | 6 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 7 | 3 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 5 | 2 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 4 | 2 | 2 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.